CLINICAL TRIAL: NCT06020157
Title: Comparison of Simple and Continuous Suture Techniques in Oral Surgery Regarding Wound Healing, a Split-Mouth Clinical Trial
Brief Title: Comparison of Simple and Continuous Suture Techniques in Oral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Selcuk003
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Suture Group (Experimental)
  Interventions: Other: Simple Suture Technique
- Continuous Suture Group (Experimental)
  Interventions: Other: Continuous Suture Technique

INTERVENTIONS:
Other: Simple Suture Technique — The half of the full arch flap will be closed by the simple suture technique.
  Arms: Simple Suture Group
Other: Continuous Suture Technique — The half of the full arch flap will be closed by the continuous suture technique.
  Arms: Continuous Suture Group

SUMMARY:
The study aims to compare two different suture techniques regarding wound healing. In this research, which is designed as a prospective study, a comparison of simple and locked continuous suture techniques will be done. For this purpose, Selçuk University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, being treated at the full arch flap opened (for alveoplasty). Half of the arch will be closed by a simple suture. The other half will be closed by continuous suture technique.

It is planned to evaluate wound healing with the Landry Healing Index and Early Wound Healing Score. It is planned to measure the amount of knot looseness in millimeters on the 7th day when the sutures will be removed. On the 7th day, it is planned to evaluate the suture removal pain for the patient and the ease of suture removal for the operator with the VAS scale. Data collected from these assessments will be statistically compared for simple and continuous sutures.

ELIGIBILITY:
Inclusion Criteria:

* Needing full arch alveoplasty
* No smoking

Exclusion Criteria:

* Uncontrolled systemic condition
* Not participating in control appointments
* Complications about wound healing

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Early Wound Healing Score-1 | Day 1
  Scoring wound healing according to Early Wound Healing Score(1 to 10; 1 is the best/10 is the worst)
Early Wound Healing Score-3 | Day 3
  Scoring wound healing according to Early Wound Healing Score(1 to 10; 1 is the best/10 is the worst)
Early Wound Healing Score-7 | Day 7
  Scoring wound healing according to Early Wound Healing Score(1 to 10; 1 is the best/10 is the worst)
Suturing Time | 1 minutes after ending suture
  The time between start and end of suture
Pain at Suture Removal | Day 7
  VAS scoring for pain at suture removal. The range of Scala is 0-10. A lower score means better results.
Suture Removal Difficulty | Day 7
  VAS scoring for suture removal difficulty. The range of Scala is 0-10. A lower score means better results.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Koyuncu, Principal Investigator — Selcuk University, Faculty of Dentistry
Locations (1):
- Selcuk University, Dentistry Faculty, Konya, Selçuklu, Turkey (Türkiye)